CLINICAL TRIAL: NCT06121999
Title: 13-Week Behavioral Lifestyle Intervention for Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) and Metabolic Dysfunction-associated Steatosis (MASH) in Adults: A Randomized Control Trial
Brief Title: Behavioral Lifestyle Intervention for Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Collaborators: Gastroenterology Associates of Western Michigan (Unknown)
Responsible Party: Principal Investigator, Scott Truskowski, OST Department Chair, Associate Professor Occupational Science and Therapy Department, Grand Valley State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-278-H
Record Dates: First submitted 2023-09-28; First posted 2023-11-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Associated-dysfunction Steatotic Liver Disease (MASLD); Metabolic Associated-dysfunction Steatohepatitis (MASH)
Keywords: weight loss; lifestyle modification; behavior change; liver disease; physical activity; nonalcoholic fatty liver disease (NAFLD); nonalcoholic steatohepatitis (NASH); noncommunicable disease; chronic disease; obesity
MeSH Terms: conditions — Weight Loss; Liver Diseases; Motor Activity; Non-alcoholic Fatty Liver Disease; Noncommunicable Diseases; Chronic Disease; Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the control or experimental intervention on a rolling basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance-based behavioral weight loss program (ABWL) (Active Comparator): Participants meet individually for 30 - 60 minutes with an occupational therapist for 13 consecutive weeks at a gastroenterology office. Outcome data is collected at baseline (visit 1) and at the end of the study (visit 13), Participants work on two modules per week in-between visits. During visits the participants' weight is recorded, module contents and worksheet information is reviewed and recorded, and suggestions are made as indicated in the clinician guide.
  Interventions: Behavioral: Standard of care acceptance-based behavioral weight loss program
- Occupational Therapy behavioral lifestyle intervention (Experimental): Participants meet individually for 60-90 minutes with an occupational therapist for 13 consecutive weeks at a gastroenterology office. Outcome data is collected at baseline (visit 1) and at the end of the study (visit 13). The Model of Human Occupation Screening Tool (MOHOST) and Role Checklist version 3 (RCv3) assessment are also used for intervention in the areas of motivation for occupation, pattern of occupation, communication & interaction skills, motor skills, process skills, and environment. Participants are also educated about practice guidelines for MASLD/MASH such as a Mediterranean (MED) diet and a personalized exercise plan. In-between visits, participants work on two modules of the control intervention and implement dietary and lifestyle modifications discussed during the visit.
  Interventions: Behavioral: Standard of care acceptance-based behavioral weight loss program; Behavioral: Occupational therapy dietary and lifestyle modifications

INTERVENTIONS:
Behavioral: Standard of care acceptance-based behavioral weight loss program — Evidence-based, structured weight loss program for adults with co-morbid conditions of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH). Published as a workbook for participants and a clinician guide, the intervention consists of twenty-five sessions or modules with accompanying worksheets. Each session covers specific acceptance-based behavioral skills to implement and build upon in subsequent sessions.
Behavioral: Occupational therapy dietary and lifestyle modifications — Occupational therapy Model of Human Occupation Screening Tool (MOHOST) and Role Checklist version 3 (RCv3) assessments identify areas of need for personalizing participant implementation of the standard of care acceptance-based behavioral weight loss program. Areas of need may include physical activity limitations to be addressed in an exercise plan or social determinants of health that are barriers to dietary and lifestyle modifications. Dietary and lifestyle modifications are based on American Gastroenterology Association (AGA) recommendations published in practice guidelines for this population. Recommendations include a Mediterranean diet, improved self-management of co-morbid chronic conditions, and a total body weight loss of five to ten percent at 1 - 2 pound weekly increments.
  Arms: Occupational Therapy behavioral lifestyle intervention

SUMMARY:
The goal of this randomized control trial study is to compare an acceptance-based weight loss program with an occupational therapy behavioral lifestyle modification intervention in adults with metabolic associated-dysfunction steatotic liver disease (MASLD) and metabolic associated-dysfunction steatohepatitis (MASH). Formerly known as nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH). The main questions the study aims to answer are:

1. How do the two interventions compare for improving weight loss, health-related quality of life (HRQOL), and FibroScan results.
2. Examine the role of occupational therapy on a multidisciplinary team for the treatment of MASLD and MASH.

Participants will meet with an occupational therapist for individual, 60-minute visits for 13 consecutive weeks. Each week participants will be weighed and then engage in a personalized intervention. At the end of the visit participants will be given worksheets and information to work on in-between visits.

Researchers will compare the intervention with an acceptance-based behavioral weight loss program that is commonly used for people with obesity and or type 2 diabetes.

DETAILED DESCRIPTION:
The research design is a pretest-posttest randomized control trial. Forty participants will be enrolled on a rolling bases and then assigned to one of two interventions. Occupational therapy with an acceptance-based behavioral weight loss program or only the acceptance-based behavioral weight loss program. Participants for both interventions will meet with an occupational therapist individually for 60 minutes for 13 consecutive weeks. Participants will be given modules from the weight loss program and worksheets to work on in-between sessions. Individuals in the occupational therapy intervention will also work on creating and individualized physical activity plan and implementation of the Mediterranean or Med Diet. At the beginning of each visit, participants will be weighed. During the visit their food logs and worksheets will be reviewed with the participant. Additional measurements during the 1st, 7th, and 13th visit include a liver FibroScan, waist measurement, and completion of questionnaires and assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with NAFLD or NASH and have a body mass index greater than 25
* Able to provide written and verbal consent to participate in the study
* Live in the community and able their health status is such that they can be seen in the gastroenterology clinical practice
* Must be patients of Gastroenterology Associates of Western Michigan.

Exclusion Criteria:

* diagnoses or the presence of other chronic liver and biliary diseases
* enrolled in a clinical trial for NAFLD or NASH
* Completed bariatric surgery less than 12-months prior to the start of the study
* Achieved a 5% or greater total body weight loss within 6-months of the start of the study.
* Presence of significant medical or psychiatric condition

  _ Presence of cognitive impairments that would inhibit participation in the study
* Individuals who are nursing, pregnant, or planning on becoming pregnant during the study.
* Individuals with a high likelihood of loss to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
The mean % of total body weight loss (%TBWL) | End of study, week 13
  The mean % of total body weight loss (%TBWL) measures the average percentage of total body weight loss (%TBWL). Possible scores range from 1 to 15%, with higher scores indicating a better outcome.
The percentage of participants achieving a greater than or equal to 5% total body weight loss (TBWL). | End of study, week 13
  The percentage of participants achieving a greater than or equal to 5% total body weight loss (TBWL) measures the proportion of participants who achieved the weight loss goal. Possible scores range from 1 - 100%, with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Mean change in the Chronic Liver Disease Questionnaire - NAFLD/NASH (CLDQ-NAFLD/NASH) | Baseline, week 1 compared to end of study, week 13
  The mean change of the CLDQ-NAFLD / NASH measures the average in the score of the instrument. The CLDQ-NAFLD / NASH questionnaire is an evidence-based, liver specific instrument responsive to changes in health related quality of life (HRQL). Thirty-six questions measure quality of life and the health burden related to nonalcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH). Scores can range from 36-252, with higher scores indicating a better outcome.
Mean change in the kilopascals (kPa) and controlled attenuation pattern in decibels per meter (CAP dB/m) liver FibroScan scores | Baseline, week 1 compared to end of study, week 13
  The mean change of liver steatosis is measured as a controlled attenuation pattern in decibels per meter (CAP dB/m). Liver fibrosis measured as kilopascals (kPa). FibroScan liver elastography is an evidence-based, liver specific instrument that is responses to changes in liver fat (steatosis) and liver stiffness (fibrosis). The CAP dB/m score will range from 100 dB/m to 400 dB/m with lower scores indicating a better outcome. The kPA score will range from 2 kPa to 14 kPA (for non-cirrhotic patients) with lower scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Truskowski, PhD, Principal Investigator — Grand Valley State University
Locations (1):
- Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant identification information will be de-identified. The de-identified data will be shared.

REFERENCES:
- [Background] Forman EM, Butryn ML. A new look at the science of weight control: how acceptance and commitment strategies can address the challenge of self-regulation. Appetite. 2015 Jan;84:171-80. doi: 10.1016/j.appet.2014.10.004. Epub 2014 Oct 16. PMID 25445199
- [Background] Gu Y, Zhou R, Kong T, Zhang W, Chen Y, Wang C, Shi J, Hu Y. Barriers and enabling factors in weight management of patients with nonalcoholic fatty liver disease: A qualitative study using the COM-B model of behaviour. Health Expect. 2023 Feb;26(1):355-365. doi: 10.1111/hex.13665. Epub 2022 Nov 16. PMID 36385729
- [Background] Kanwal F, Shubrook JH, Younossi Z, Natarajan Y, Bugianesi E, Rinella ME, Harrison SA, Mantzoros C, Pfotenhauer K, Klein S, Eckel RH, Kruger D, El-Serag H, Cusi K. Preparing for the NASH Epidemic: A Call to Action. Gastroenterology. 2021 Sep;161(3):1030-1042.e8. doi: 10.1053/j.gastro.2021.04.074. Epub 2021 Jul 26. PMID 34416976
- [Background] Kanwal F, Shubrook JH, Adams LA, Pfotenhauer K, Wai-Sun Wong V, Wright E, Abdelmalek MF, Harrison SA, Loomba R, Mantzoros CS, Bugianesi E, Eckel RH, Kaplan LM, El-Serag HB, Cusi K. Clinical Care Pathway for the Risk Stratification and Management of Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2021 Nov;161(5):1657-1669. doi: 10.1053/j.gastro.2021.07.049. Epub 2021 Sep 20. PMID 34602251
- [Background] Konerman MA, Walden P, Joseph M, Jackson EA, Lok AS, Rubenfire M. Impact of a structured lifestyle programme on patients with metabolic syndrome complicated by non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2019 Feb;49(3):296-307. doi: 10.1111/apt.15063. Epub 2018 Dec 18. PMID 30561027
- [Background] Ng CH, Lim WH, Chin YH, Yong JN, Zeng RW, Chan KE, Tan DJH, Fu CE, Tang ASP, Goh LH, Devi K, Chew NWS, Mak LL, Tamaki N, Huang DQ, Noureddin M, Siddiqui MS, Loomba R, Sanyal AJ, Muthiah M. Living in the non-alcoholic fatty liver disease silent epidemic: a qualitative systematic review of patients' perspectives. Aliment Pharmacol Ther. 2022 Aug;56(4):570-579. doi: 10.1111/apt.17121. Epub 2022 Jul 6. PMID 35791632
- [Background] Scott PJ. Occupational therapy services to enable liver patients to thrive following transplantation. Occup Ther Health Care. 2011 Oct;25(4):240-56. doi: 10.3109/07380577.2011.600427. Epub 2011 Aug 9. PMID 23899078
- [Background] Scott PJ, Brown VL. Resumption of valued activities in the first year post liver transplant. Occup Ther Health Care. 2012 Jan;26(1):48-63. doi: 10.3109/07380577.2011.643856. PMID 23899107
- [Background] Arshad T, Henry L, Younossi ZM. Validation of the chronic liver disease questionnaire for non-alcoholic steatohepatitis in patients: impact for the clinic. Expert Rev Gastroenterol Hepatol. 2019 Aug;13(8):709-710. doi: 10.1080/17474124.2019.1636646. Epub 2019 Jun 28. No abstract available. PMID 31248299
- [Background] Bahadir Agce Z, Ekici G. Person-centred, occupation-based intervention program supported with problem-solving therapy for type 2 diabetes: a randomized controlled trial. Health Qual Life Outcomes. 2020 Aug 3;18(1):265. doi: 10.1186/s12955-020-01521-x. PMID 32746841
- [Background] Younossi ZM, Corey KE, Lim JK. AGA Clinical Practice Update on Lifestyle Modification Using Diet and Exercise to Achieve Weight Loss in the Management of Nonalcoholic Fatty Liver Disease: Expert Review. Gastroenterology. 2021 Feb;160(3):912-918. doi: 10.1053/j.gastro.2020.11.051. Epub 2020 Dec 9. PMID 33307021
- [Background] Younossi ZM, Stepanova M, Younossi I, Racila A. Validation of Chronic Liver Disease Questionnaire for Nonalcoholic Steatohepatitis in Patients With Biopsy-Proven Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2093-2100.e3. doi: 10.1016/j.cgh.2019.01.001. Epub 2019 Jan 11. PMID 30639779
- [Background] Scott PJ, McKinney KG, Perron JM, Ruff EG, Smiley JL. The Revised Role Checklist: Improved Utility, Feasibility, and Reliability. OTJR (Thorofare N J). 2019 Jan;39(1):56-63. doi: 10.1177/1539449218780618. Epub 2018 Jun 20. PMID 29923446
- [Background] Occupational Therapy Practice Framework: Domain and Process-Fourth Edition. Am J Occup Ther. 2020 Aug 1;74(Supplement_2):7412410010p1-7412410010p87. doi: 10.5014/ajot.2020.74S2001. PMID 34780625
- [Background] Bischoff M, Zimny S, Feiner S, Sauter J, Sydor S, Denk G, Nagel JM, Bischoff G, Rust C, Hohenester S. Multidisciplinary lifestyle intervention is associated with improvements in liver damage and in surrogate scores of NAFLD and liver fibrosis in morbidly obese patients. Eur J Nutr. 2022 Aug;61(5):2725-2735. doi: 10.1007/s00394-022-02846-7. Epub 2022 Mar 11. PMID 35277756
- [Background] Buzzetti E, Linden A, Best LM, Madden AM, Roberts D, Chase TJG, Freeman SC, Cooper NJ, Sutton AJ, Fritche D, Milne EJ, Wright K, Pavlov CS, Davidson BR, Tsochatzis E, Gurusamy KS. Lifestyle modifications for nonalcohol-related fatty liver disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 11;6(6):CD013156. doi: 10.1002/14651858.CD013156.pub2. PMID 34114650
- [Background] Chan WK, Chuah KH, Rajaram RB, Lim LL, Ratnasingam J, Vethakkan SR. Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): A State-of-the-Art Review. J Obes Metab Syndr. 2023 Sep 30;32(3):197-213. doi: 10.7570/jomes23052. Epub 2023 Sep 13. PMID 37700494
- [Background] Chai XN, Zhou BQ, Ning N, Pan T, Xu F, He SH, Chen NN, Sun M. Effects of lifestyle intervention on adults with metabolic associated fatty liver disease: A systematic review and meta-analysis. Front Endocrinol (Lausanne). 2023 Feb 16;14:1081096. doi: 10.3389/fendo.2023.1081096. eCollection 2023. PMID 36875459
- [Background] Cook NS, Nagar SH, Jain A, Balp MM, Maylander M, Weiss O, Chatterjee S. Understanding Patient Preferences and Unmet Needs in Non-alcoholic Steatohepatitis (NASH): Insights from a Qualitative Online Bulletin Board Study. Adv Ther. 2019 Feb;36(2):478-491. doi: 10.1007/s12325-018-0856-0. Epub 2018 Dec 13. PMID 30547371
- [Background] Dhaliwal HS, Singh R, Abraham AM, Sharma R, Goyal NK, Soloman R, Bansal P, Goyal A. Perception of Illness and Its Association with Treatment Willingness in Patients with Newly Diagnosed Nonalcoholic Fatty Liver Disease. Dig Dis Sci. 2021 Dec;66(12):4197-4207. doi: 10.1007/s10620-020-06794-2. Epub 2021 Jan 6. PMID 33409801
- [Background] Fields B, Smallfield S. Occupational Therapy Practice Guidelines for Adults With Chronic Conditions. Am J Occup Ther. 2022 Mar 1;76(2):7602397010. doi: 10.5014/ajot.2022/762001. PMID 35311934
- [Background] Glass L, Asefa H, Volk M, Lok AS, Tincopa MA. Disease Knowledge, Health-Related Quality of Life, and Lifestyle Behavior Change in Patients with Nonalcoholic Fatty Liver Disease: Impact of an Educational Intervention. Dig Dis Sci. 2022 Jun;67(6):2123-2133. doi: 10.1007/s10620-021-07052-9. Epub 2021 May 27. PMID 34043121
- [Background] Glass O, Liu D, Bechard E, Guy CD, Pendergast J, Mae Diehl A, Abdelmalek MF. Perceptions of Exercise and Its Challenges in Patients With Nonalcoholic Fatty Liver Disease: A Survey-Based Study. Hepatol Commun. 2022 Feb;6(2):334-344. doi: 10.1002/hep4.1808. Epub 2021 Oct 26. PMID 34697917
- [Background] Heredia NI, Gaba R, Liu Y, Jain S, Rungta M, Rungta M, El-Serag HB, Kanwal F, Thrift AP, Balakrishnan M. Perceptions of weight status and energy balance behaviors among patients with non-alcoholic fatty liver disease. Sci Rep. 2022 Apr 5;12(1):5695. doi: 10.1038/s41598-022-09583-1. PMID 35383229
- [Background] Hershman M, Torbjornsen K, Pang D, Wyatt B, Dieterich DT, Perumalswami PV, Branch AD, Dinani AM. Modification of the diabetes prevention program for the treatment of nonalcoholic fatty liver disease: A pilot study. Obes Sci Pract. 2022 Oct 20;9(3):218-225. doi: 10.1002/osp4.637. eCollection 2023 Jun. PMID 37287520
- [Background] Balakrishnan M, Liu K, Schmitt S, Heredia NI, Sisson A, Montealegre JR, Hernaez R, Kanwal F, Foreyt J. Behavioral weight-loss interventions for patients with NAFLD: A systematic scoping review. Hepatol Commun. 2023 Aug 3;7(8):e0224. doi: 10.1097/HC9.0000000000000224. eCollection 2023 Aug 1. PMID 37534947
- [Background] Keating SE, Sabag A, Hallsworth K, Hickman IJ, Macdonald GA, Stine JG, George J, Johnson NA. Exercise in the Management of Metabolic-Associated Fatty Liver Disease (MAFLD) in Adults: A Position Statement from Exercise and Sport Science Australia. Sports Med. 2023 Dec;53(12):2347-2371. doi: 10.1007/s40279-023-01918-w. Epub 2023 Sep 11. PMID 37695493
- [Background] Park J, Gross DP, Rayani F, Norris CM, Roberts MR, James C, Guptill C, Esmail S. Model of Human Occupation as a framework for implementation of Motivational Interviewing in occupational rehabilitation. Work. 2019;62(4):629-641. doi: 10.3233/WOR-192895. PMID 31104046
- [Background] Ho ECM, Siu AMH. Occupational Therapy Practice in Sleep Management: A Review of Conceptual Models and Research Evidence. Occup Ther Int. 2018 Jul 29;2018:8637498. doi: 10.1155/2018/8637498. eCollection 2018. PMID 30150906
- [Background] Mack RA, Stanton CE, Carney MR. The importance of including occupational therapists as part of the multidisciplinary team in the management of eating disorders: a narrative review incorporating lived experience. J Eat Disord. 2023 Mar 9;11(1):37. doi: 10.1186/s40337-023-00763-6. PMID 36894981
- [Background] Edgelow MM, MacPherson MM, Arnaly F, Tam-Seto L, Cramm HA. Occupational therapy and posttraumatic stress disorder: A scoping review. Can J Occup Ther. 2019 Apr;86(2):148-157. doi: 10.1177/0008417419831438. Epub 2019 Apr 23. PMID 31014080
- [Background] Goodman V, Wardrope B, Myers S, Cohen S, McCorquodale L, Kinsella EA. Mindfulness and human occupation: A scoping review. Scand J Occup Ther. 2019 Apr;26(3):157-170. doi: 10.1080/11038128.2018.1483422. Epub 2018 Jun 28. PMID 29952233
- [Background] Nielsen SS, Skou ST, Larsen AE, Polianskis R, Pawlak WZ, Vaegter HB, Sondergaard J, Christensen JR. Occupational therapy lifestyle intervention added to multidisciplinary treatment for adults living with chronic pain: a feasibility study. BMJ Open. 2022 Sep 17;12(9):e060920. doi: 10.1136/bmjopen-2022-060920. PMID 36115674
- [Background] Meidert U, Bonsaksen T, Scott PJ. A study of measuring participation according to the International Classification of Functioning, Disability and Health with the Revised Role Checklist. Clin Rehabil. 2018 Nov;32(11):1530-1539. doi: 10.1177/0269215518782339. Epub 2018 Jun 25. PMID 29938529
- [Background] Mobasheri N, Ghahremani L, Fallahzadeh Abarghooee E, Hassanzadeh J. Lifestyle Intervention for Patients with Nonalcoholic Fatty Liver Disease: A Randomized Clinical Trial Based on the Theory of Planned Behavior. Biomed Res Int. 2022 Sep 12;2022:3465980. doi: 10.1155/2022/3465980. eCollection 2022. PMID 36132088
- [Background] Rinella ME, Neuschwander-Tetri BA, Siddiqui MS, Abdelmalek MF, Caldwell S, Barb D, Kleiner DE, Loomba R. AASLD Practice Guidance on the clinical assessment and management of nonalcoholic fatty liver disease. Hepatology. 2023 May 1;77(5):1797-1835. doi: 10.1097/HEP.0000000000000323. Epub 2023 Mar 17. No abstract available. PMID 36727674
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Castro Narro GE, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. Hepatology. 2023 Dec 1;78(6):1966-1986. doi: 10.1097/HEP.0000000000000520. Epub 2023 Jun 24. PMID 37363821
- [Background] Romero-Gomez M, Zelber-Sagi S, Trenell M. Treatment of NAFLD with diet, physical activity and exercise. J Hepatol. 2017 Oct;67(4):829-846. doi: 10.1016/j.jhep.2017.05.016. Epub 2017 May 23. PMID 28545937
- [Background] Smallfield S, Fang L, Kyler D. Self-Management Interventions to Improve Activities of Daily Living and Rest and Sleep for Adults With Chronic Conditions: A Systematic Review. Am J Occup Ther. 2021 Jul 1;75(4):7504190010. doi: 10.5014/ajot.2021.046946. PMID 34780611
- [Background] Tomah S, Salah T, Al-Badri M, Dhaver S, Gardner H, Tasabehji MW, Hamdy O. Multidisciplinary intensive lifestyle intervention improves markers of nonalcoholic fatty liver disease (NAFLD) in patients with type 1 diabetes and obesity: a retrospective matched-cohort study. Clin Diabetes Endocrinol. 2023 Apr 12;9(1):3. doi: 10.1186/s40842-023-00150-9. PMID 37046323
- [Background] Wang L, Zhou H, Liu Y, Wang X, Yan W, Zhang J, Ren H. Factors influencing adherence to lifestyle prescriptions among patients with nonalcoholic fatty liver disease: A qualitative study using the health action process approach framework. Front Public Health. 2023 Mar 17;11:1131827. doi: 10.3389/fpubh.2023.1131827. eCollection 2023. PMID 37006574
- [Background] Younossi ZM, Zelber-Sagi S, Henry L, Gerber LH. Lifestyle interventions in nonalcoholic fatty liver disease. Nat Rev Gastroenterol Hepatol. 2023 Nov;20(11):708-722. doi: 10.1038/s41575-023-00800-4. Epub 2023 Jul 4. PMID 37402873
- [Background] Younossi ZM, Stepanova M, Henry L, Racila A, Lam B, Pham HT, Hunt S. A disease-specific quality of life instrument for non-alcoholic fatty liver disease and non-alcoholic steatohepatitis: CLDQ-NAFLD. Liver Int. 2017 Aug;37(8):1209-1218. doi: 10.1111/liv.13391. Epub 2017 Mar 13. PMID 28211165